CLINICAL TRIAL: NCT01214668
Title: A Phase 1b, Multicenter, Dose-Escalation Study of LY573636-sodium in Combination With Liposomal Doxorubicin in Patients With Advanced Solid Tumors
Brief Title: Dose-Escalation Study of LY573636-sodium and Liposomal Doxorubicin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12887; H8K-MC-JZAN (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY573636 + Liposomal Doxorubicin (Experimental)
  Interventions: Drug: LY573636-sodium; Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: LY573636-sodium — Individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28-day cycle.
  Participants may continue on study drug until disease progression, unacceptable toxicity, cumulative dose of 550 milligrams per square meter (mg/m²) of liposomal doxorubicin or doxorubicin is reached, or other withdrawal criterion is met.
  Other Names: Tasisulam-sodium
Drug: Liposomal Doxorubicin — 40 mg/m² on Day 1, given intravenously of each 28-day cycle
  Participants may continue on study drug until disease progression, unacceptable toxicity, cumulative dose of 550 mg/m² of liposomal doxorubicin or doxorubicin is reached, or other withdrawal criterion are met.

SUMMARY:
The goal of this study is to determine the dose of LY573636-sodium (hereafter referred to as LY573636) that can be administered safely in combination with liposomal doxorubicin in patients with advanced cancer who have failed a prior treatment.

The study consists of a dose escalation phase to the maximum tolerated dose (MTD) and a dose confirmation phase in patients with platinum resistant epithelial ovarian, fallopian tube or primary peritoneal cancer who have never been treated with doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* You must have a histologically confirmed solid malignancy that is unresectable and/or metastatic which has progressed after receiving standard approved chemotherapy
* You must have a solid malignancy for which an anthracycline-based regimen is felt to be a reasonable treatment option
* You must have measurable disease or non-measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
* You must have a serum albumin level greater than or equal to 3.0 grams/deciliter (g/dL) (30 g/L)
* You must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* You must have tumor progression after receiving standard/approved chemotherapy
* You must be reliable and willing to make yourself available for the duration of the study and are willing to follow study procedures
* Women must be sterile, post-menopausal or on a contraception and men must be sterile or on contraception
* Your test results assessing the function of your blood, kidneys, liver, and heart are satisfactory
* Ovarian patients in the confirmation phase must have failed to achieve at least a partial response to a first-line platinum-based therapy (platinum-refractory) or have progression in less than 6 months after a response to a first-line platinum-based therapy (platinum-resistant)
* Ovarian patients in the confirmation phase must have measurable disease by RECIST
* Ovarian patients in the confirmation phase must be liposomal doxorubicin or doxorubicin naive and not amendable to curative therapy

Exclusion Criteria:

* You cannot have received other investigational drugs within the last 28 days
* You cannot have other on-going serious illnesses including active bacterial, fugal, or viral infections
* You cannot have current hematologic malignancies, acute or chronic leukemia, or brain metastasis
* You cannot currently be receiving warfarin (Coumadin®) therapy
* You cannot have known positive test results in human immunodeficiency, hepatitis B surface antigen or hepatitis C antibodies
* You cannot have a history of cardiac disease or clinical evidence of congestive heart failure
* Ovarian patients in the confirmation phase who have received 2 or more cytotoxic regimens for platinum-resistant disease
* You cannot currently be receiving amiodarone, quinidine, propofol, and clozapine
* If you are taking esomeprazole or pantoprazole you must be able to stop taking this medication within 72 hours before and after LY573636 administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-651-4559 Mon. - Fri. 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Encinitas, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment and a participant was considered to have "completed" the trial if they experienced progressive disease or an adverse event.
Groups:
- LY 300 μg/mL + Dox: LY573636 targeting a maximum concentration (Cmax) of 300 micrograms per milliliter (μg/mL) (LY 300 μg/mL) as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 milligrams per square meter (mg/m²) during the Dose-Escalation Phase.
- LY 320 μg/mL + Dox: LY573636 targeting a Cmax of 320 μg/mL (LY 320 μg/mL) as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Escalation Phase.
- LY 340 μg/mL + Dox: LY573636 targeting a Cmax of 340 μg/mL (LY 340 μg/mL) as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Escalation Phase.
- LY 360 μg/mL + Dox: LY573636 targeting a Cmax of 360 μg/mL (LY 360 μg/mL) as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Escalation Phase.
- LY 380 μg/mL + Dox: LY573636 targeting a Cmax of 380 μg/mL (LY 380 μg/mL) as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Escalation Phase.
- LY Albumin and Day 15 PK Tailored + Dox: LY573636 dosing was given as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Confirmation Phase. LY573636 dose was based on an albumin-corrected exposure (AUCalb) target range of 75th percentile of 3500 hour*micrograms per milliliter (h*µg/mL) and the Cycle 1, Day 15 LY573636 total drug level (Day 15 pharmacokinetic [PK]) (LY Albumin and Day 15 PK Tailored).
Period: Overall Study
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Started | 4 | 3 | 6 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 4 | 3 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 6 | 6 | 6 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 4 | 2 | 5 | 4 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who had at least one dose of study drug.
Groups:
- LY Albumin and Day 15 PK Tailored + Dox: LY573636 dosing was given as a 2-hour infusion on Day 1 of a 28-day cycle in combination with liposomal doxorubicin (Dox) at a dose of 40 mg/m² during the Dose-Confirmation Phase. LY573636 dose was based on an albumin-corrected exposure (AUCalb) target range of 75th percentile of 3500 hour*micrograms per milliliter (h*μg/mL) and the Cycle 1, Day 15 LY573636 total drug level (Day 15 pharmacokinetic [PK]) (LY Albumin and Day 15 PK Tailored).
- Total: Total of all reporting groups
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox | Total
Number analyzed (Participants) | 4 | 3 | 6 | 6 | 6 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.39 (13.60) | 51.54 (8.55) | 64.65 (7.53) | 58.57 (2.71) | 52.24 (15.08) | 57.82 (12.97) | 57.54 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 5 | 5 | 6 | 28
  Male | 0 | 1 | 0 | 1 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 2 | 0 | 6
  Not Hispanic or Latino | 2 | 2 | 6 | 5 | 4 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 5 | 6 | 5 | 6 | 28
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 6 | 6 | 6 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD), which is corrected for the participant's predose albumin to identify the albumin-corrected exposure range of LY 573636 when combined with liposomal doxorubicin. MTD is the highest dose with <33% of participants having a dose-limiting toxicity (DLT) in the first 28-day cycle of treatment. DLT is an adverse event (AE) that is likely related to the study drug or combination and fulfills any 1 of the following: Common Terminology Criteria for AE (CTCAE, Version 3.0) Grade (Gr) 4 hematologic toxicity; Gr 3 nonhematologic toxicity (excluding controllable nausea/vomiting or diarrhea and alopecia); Gr 3 electrolyte toxicity that is not resolved with standard treatments. Those who enter the study with Gr 2 hepatic enzyme abnormalities, DLT for an isolated Gr 3 hepatic enzyme abnormality is determined by investigators; a DLT can be declared if a participant experiences increasing toxicity during treatment.
Time Frame: Predose up to 28 days postdose in Cycle 1
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: micrograms per milliliter (μg/mL)
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Number analyzed (Participants) | 4 | 3 | 6 | 6 | 6 | 6
micrograms per milliliter (μg/mL) | NA — MTD was not reached because none of the participants reached the criteria for MTD. | NA — MTD was not reached because none of the participants reached the criteria for MTD. | NA — MTD was not reached because none of the participants reached the criteria for MTD. | NA — MTD was not reached because none of the participants reached the criteria for MTD. | NA — MTD was not reached because none of the participants reached the criteria for MTD. | NA — MTD was not reached because none of the participants reached the criteria for MTD.

2. Secondary Outcome: Number of Participants With Clinically Significant Events
Description: Clinically significant events are defined as serious adverse events (SAEs), regardless of causality, during the study including the 30-day follow-up period. A summary of SAEs and other nonserious adverse events is located in the Reported Adverse Event section. Death due to progressive disease was not considered as an SAE.
Time Frame: Baseline to study completion up to 18.49 months
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Number analyzed (Participants) | 4 | 3 | 6 | 6 | 6 | 6
Participants | 2 | 0 | 5 | 3 | 3 | 3

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY573636
Time Frame: Predose, 30 minutes (min), 2 hours (h), 4 h, 166 h, 360 h and 698 h postdose in Cycle 1; Predose, 30 min, 2 h, 4 h, 166 h, 360 h and 698 h postdose in Cycle 2; Predose, 166h, 360h and 698 h postdose in Cycle 3
Population: Participants who received the study drug and had sufficient pharmacokinetic (PK) data to estimate Cmax at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- LY573636: LY573636 dose was based on an albumin-corrected exposure (AUCalb) to target a specific exposure range. Intravenous dosing is done on Day 1 of a 28-day cycle. Data are pooled together from all treatment groups.
Arm/Group | LY573636
Number analyzed (Participants) | 31
micrograms per milliliter (µg/mL)
  Cycle 1 | 335.1 (13.9)
  Cycle 2: number analyzed (Participants) | 27
  Cycle 2 | 284.5 (15.9)
  Cycle 3: number analyzed (Participants) | 21
  Cycle 3 | 250.7 (25.2)

4. Secondary Outcome: Number of Participants With Tumor Response
Description: Number of participants with tumor response = number of participants with complete response (CR) + number of participants with partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is the disappearance of all target and non-target lesions; PR is a ≥30% decrease in the sum of longest diameter of target lesions.
Time Frame: Baseline to measured progressive disease up to 4.7 months
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Number analyzed (Participants) | 4 | 3 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 3 | 0 | 2

5. Secondary Outcome: Pharmacokinetics: Area Under the Curve of LY573636 Above the Albumin Corrected Threshold (AUCalb)
Description: LY573636 has been found to be highly bound to albumin. AUCalb is a surrogate measure of exposure to unbound (free) LY573636.
Time Frame: Predose, 30 min, 2 h, 4 h, 166 h, 360 h and 698 h postdose in Cycle 1; Predose, 30 min, 2 h, 4 h, 166 h, 360 h and 698 h postdose in Cycle 2; Predose, 166h, 360h and 698 h postdose in Cycle 3
Population: Participants who received the study drug and had sufficient pharmacokinetic (PK) data to calculate AUCalb at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter (h*µg/mL)
Arm/Group | LY573636
Number analyzed (Participants) | 31
hour*micrograms per milliliter (h*µg/mL)
  Cycle 1 | 1081.0 (163.9)
  Cycle 2: number analyzed (Participants) | 28
  Cycle 2 | 413.7 (684.3)
  Cycle 3: number analyzed (Participants) | 19
  Cycle 3 | 228.4 (323.3)

6. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease During the 30 Days Following Discontinuation From Study Treatment
Time Frame: From date of randomization until up to 30 days post study treatment discontinuation, assessed up to 4.7 months
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Number analyzed (Participants) | 4 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events and are reported in the Other Pre-Specified Outcome Measure for those who died within the 30-day post study treatment follow-up period.
Arm/Group | LY 300 μg/mL + Dox | LY 320 μg/mL + Dox | LY 340 μg/mL + Dox | LY 360 μg/mL + Dox | LY 380 μg/mL + Dox | LY Albumin and Day 15 PK Tailored + Dox
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 5/6 | 3/6 | 3/6 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 300 μg/mL + Dox (N=4) | LY 320 μg/mL + Dox (N=3) | LY 340 μg/mL + Dox (N=6) | LY 360 μg/mL + Dox (N=6) | LY 380 μg/mL + Dox (N=6) | LY Albumin and Day 15 PK Tailored + Dox (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This event resulted in death.
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 300 μg/mL + Dox (N=4) | LY 320 μg/mL + Dox (N=3) | LY 340 μg/mL + Dox (N=6) | LY 360 μg/mL + Dox (N=6) | LY 380 μg/mL + Dox (N=6) | LY Albumin and Day 15 PK Tailored + Dox (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 4 (5) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 5 (5) | 2 (2) | 1 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 3 (4)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (6) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (2) | 5 (5) | 2 (2) | 4 (5) | 2 (2)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (2) | 1 (2) | 2 (2) | 3 (4) | 3 (5) | 3 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 4 (5) | 4 (5) | 2 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 4 (6) | 3 (5) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contraceptive diaphragm (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days